CLINICAL TRIAL: NCT05347277
Title: CSF Free Kappa Light Chain for The Diagnosis of Demyelinating Disorders Taking Oligoclonal Banding Via Isoelectric Focusing Electrophoresis as Gold Standard: A Laboratory Study
Brief Title: CSF Free Kappa Light Chain for The Diagnosis of Demyelinating Disorders
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sibtain Ahmed, Assistant Professor, Aga Khan University
Other Study IDs: 2021-6714-19104.
Record Dates: First submitted 2022-04-13; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OCB positive: The pattern of oligoclonal bands in CSF is reviewed by pathologist and their findings are noted as negative for the presence of CSF OCB
  Interventions: Diagnostic Test: Kappa Free Light Chain (K-FLC)
- OCB negative: The pattern of oligoclonal bands in CSF is reviewed by pathologist and their findings are noted as positive for the presence of CSF OCB
  Interventions: Diagnostic Test: Kappa Free Light Chain (K-FLC)

INTERVENTIONS:
Diagnostic Test: Kappa Free Light Chain (K-FLC) — A biochemical test measured on CSF sample via nephelometry on Beckman Immage-800 analyzer using kits from Freelite, The Binding Site, according to the manufacturer's instructions.

SUMMARY:
Multiple sclerosis (MS) is a demyelinating disease of the central nervous system (CNS) which commonly leads to disability. The current preferred clinical laboratory test for the diagnosis is the detection of oligoclonal bands (OCBs) in the cerebrospinal fluid (CSF) by isoelectric focusing electrophoresis (IEF) followed by immunoblotting.Measuring the levels of Kappa Free Light Chain (K-FLC) in CSF has been proposed as a potential alternative to the qualitative assessment of OCBs. The aim of this study is to validate and determine the diagnostic yield of K-FLC in CSF against OCBs via IEF as gold standard.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a demyelinating disease of the central nervous system (CNS) which commonly leads to disability. It is the most common disabling neurological disease found in young adults, most commonly presenting between the ages of 20 to 40 . The current preferred clinical laboratory test for the diagnosis is the detection of oligoclonal bands (OCBs) in the cerebrospinal fluid (CSF) by isoelectric focusing electrophoresis (IEF) followed by immunoblotting. This manual technique requires paired CSF and serum specimens to be run in parallel, with a subjective visual interpretation. The multi-step method is labor intensive and costly, with an average time for analytical processing of over 3 hours. There is no standard definition of OCB amounts required for a clinically positive result. With differing approaches by varied institutions, positivity can be characterized by anything from 1 to 4 unique CSF bands, which significantly affects sensitivity and specificity of the assay. Measuring the levels of Kappa Free Light Chain (K-FLC) in CSF has been proposed as a potential alternative to the qualitative assessment of OCBs. This lab-based validation study would allow the laboratory to cut spending by reducing technologist time and eliminating expensive IEF kits. Additionally, K-FLC would replace subjective interpretation with quantitative values, overcoming the challenges associated with the performance and subjective interpretation of OCB testing. The aim of this study is to validate and determine the diagnostic yield of K-FLC in CSF against OCBs via IEF as gold standard.

OCB via IEF is routinely performed at the Section of Chemical Pathology for patients with suspicion of MS or demyelinating disorders. Paired patient CSF and serum specimens are collected. The oligoclonal bands are tested by IEF on agarose gel using Interlab diagnostics CSF IEF kit and manual immunoblotting steps to transfer the proteins on transfer membranes. Simultaneous analysis is also conducted on serum samples. The pattern of oligoclonal bands in CSF is reviewed by pathologist and their findings are noted as positive or negative for presence or absence of CSF OCB or matching, that is, bands present in both serum and CSF.

The samples received during the last 3 months from June to August for OCBS via IEF are saved in the lab in frozen conditions, stable for analysis. 0.5 ml CSF sample will be utilized for analysis by nephelometry on Beckman Immage-800 analyzer using kits from Freelite, The Binding Site, according to the manufacturer's instructions.

To ensure confidentiality, all identification details will be anonymized, and study identifiers will be allotted. Additionally, all data will be stored in a password protected electronic format by the PI.

Keeping in view the low anticipated frequency of demyelinating disorders at a single center; and to achieve significant power and reliability of statistical analysis, a minimum sample size of 60 CSF samples for K-FLC analysis will be included with stratification into 3 groups: Positive (n=20), negative (n=20) and matching (n=20), for OCBs.

Data analysis will be done on SPSS version 25. Shapiro Wilk test will be used to check normality of data. Diagnostic accuracy of CSF K-FLC will be calculated on the basis of sensitivity, specificity, PPV and NPV taking OCB as gold standard. For further analysis, Receiver operative characteristic (ROC) curve will be plotted for OCB and area under the curve (AUC) will be calculated and optimal cut-off will be generated using Youden's Index. For the validation agreement between CSF L-FLC and IEF will be assessed by Cohen's kappa statistics.

ELIGIBILITY:
Inclusion Criteria:

Saved residual CSF samples positive for OCBs Saved residual CSF samples negative for OCBs

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with suspicion of MS or demyelinating disorders, routinely referred for OCBs determination via IEF at our laboratory
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Kappa Free Light Chain (KFLC) levels greater than 1 mg/L | August 2021 to August 2022
  KFLC levels greater than 1mg/L will be considered as positive for demyelinating disorders
Kappa Free Light Chain (KFLC) levels less than 1 mg/L | August 2021 to August 2022
  KFLC levels less than 1mg/L will be considered as negative for demyelinating disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Chemistry, Sopari wala building, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No